CLINICAL TRIAL: NCT02066064
Title: G-Eye Advanced Colonoscopy For Increased Polyp Detection Rate - Randomized Tandem Study With Different Endoscopist
Brief Title: G-Eye Advanced Colonoscopy For Increased Polyp Detection Rate-randomized Tandem Study With Different Endoscopist
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Smart Medical Systems Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: G-EYE
Record Dates: First submitted 2014-02-10; First posted 2014-02-19 (Estimated); Last update posted 2016-02-12 (Estimated); Status verified 2016-02

CONDITIONS: Colorectal Cancer; Adenoma
Keywords: Colorectal Cancer; Adenoma; Standard Colonoscopy; G-EYE(TM) Colonoscopy
MeSH Terms: conditions — Colorectal Neoplasms; Adenoma | interventions — Colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): Subjects will undergo complete standard colonoscopy, followed by G-EYE(TM) Colonoscopy
  Interventions: Procedure: Standard Colonoscopy; Procedure: G-EYE(TM) Colonoscopy
- Group B (Active Comparator): Subject will undergo G-EYE(TM) colonoscopy followed by standard colonoscopy
  Interventions: Procedure: Standard Colonoscopy; Procedure: G-EYE(TM) Colonoscopy

INTERVENTIONS:
Procedure: Standard Colonoscopy — Standard Colonoscopy
Procedure: G-EYE(TM) Colonoscopy — G-EYE(TM) Colonoscopy

SUMMARY:
The purpose of this study is to compare the adenoma detection rate of G-EYE™ high definition colonoscopy with that of standard high definition colonoscopy.

DETAILED DESCRIPTION:
Single Center, two-arm, randomized , open-label study with different and blinded endoscopists.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 50 years old
2. Referred to colonoscopy for screening, following positive FOBT testing, change of bowel habits or for surveillance colonoscopy (history of adenoma resection).
3. The patient must understand and provide written consent for the procedure.

Exclusion Criteria:

1. Subjects with inflammatory bowel disease;
2. Subjects with a personal history of polyposis syndrome;
3. Subjects with suspected chronic stricture potentially precluding complete colonoscopy;
4. Subjects with diverticulitis or toxic megacolon;
5. Subjects with a history of radiation therapy to abdomen or pelvis;
6. Pregnant or lactating female subjects;
7. Subjects who are currently enrolled in another clinical investigation.
8. Subjects with current oral or parenteral use of anticoagulants
9. Subjects with recent (within the last 3 mounts) coronary ischemia or CVA (stroke)

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2013-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
G-EYE™ colonoscopy detection rate of adenomas and serrated lesions compared to the standard colonoscopy detection rate of the same. | estimated 14 days (following histology results)

SECONDARY OUTCOMES:
polyp and adenoma detection, procedure times and safety | 24-72 hours post procedure

CONTACTS AND LOCATIONS:
Overall Officials: Ralf Kiesslich, Prof., Principal Investigator
Locations (1):
- St. Marienkrankenhaus Frankfurt, Frankfurt, Germany